CLINICAL TRIAL: NCT00354484
Title: Safety and Efficacy of a Hematinic Agent in the Treatment of Postpartum Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT06011
Record Dates: First submitted 2006-07-13; First posted 2006-07-20 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Postpartum Anemia
Keywords: anemia; postpartum
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): Up to a maximum cumulative dose of 2,500 mg administered IV based on iron-deficit calculations; the calculated dose was given in divided doses of up to 1,000 mg weekly.
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Ferrous Sulfate tablets (Active Comparator): 325 mg of ferrous sulfate 3 times daily (TID) x 6 weeks.
  Interventions: Drug: Ferrous Sulfate tablets

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — Up to a maximum cumulative dose of 2,500 mg administered IV based on iron-deficit calculations; the calculated dose was given in divided doses of up to 1,000 mg weekly.
  Arms: Ferric Carboxymaltose (FCM)
Drug: Ferrous Sulfate tablets — 325 mg of ferrous sulfate 3 times daily (TID) x 6 weeks.
  Arms: Ferrous Sulfate tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of VIT45 compared to the current standard of care in postpartum patients.

DETAILED DESCRIPTION:
This is an open label Phase III randomized active control study of postpartum patients with anemia. Patients will be randomized to either active control or the investigational agent and followed for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects able to give consent
* Post partum patients
* Baseline Hgb < /= 10 g/dL
* Agree to practice birth control

Exclusion Criteria:

* Participation in previous clinical trial of this investigational agent
* Known hypersensitivity reaction to active control
* Significant vaginal bleeding
* History of anemia other than iron deficiency anemia
* Anticipated need for surgery during the study
* Active severe infection or malignancy
* Known positive Hepatitis B antigen of Hepatitis C viral antibody
* Known HIV antibodies
* Received an investigational drug within 30 days of screening
* Alcohol abuse within past 6 months
* Hemochromatosis or other iron storage disorders
* Significant cardiovascular disease
* Any laboratory abnormality, medical condition or severe psychiatric disorder which in the opinion of the investigator woud put the subject's disease management at risk or may result in the subject being able to comply with the study requirements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

REFERENCES:
- [Result] Van Wyck DB, Martens MG, Seid MH, Baker JB, Mangione A. Intravenous ferric carboxymaltose compared with oral iron in the treatment of postpartum anemia: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):267-78. doi: 10.1097/01.AOG.0000275286.03283.18. PMID 17666600
- [Result] Seid MH, Rogers R, Dinh Q. Treating Postpartum Anemia with Intravenous Ferric Carboxymaltose: A Randomized Controlled Study. Southern Medical Association Scientific Assembly 2008.
- [Result] Seid MH, Derman RJ, Baker JB, Banach W, Goldberg C, Rogers R. Ferric carboxymaltose injection in the treatment of postpartum iron deficiency anemia: a randomized controlled clinical trial. Am J Obstet Gynecol. 2008 Oct;199(4):435.e1-7. doi: 10.1016/j.ajog.2008.07.046. PMID 18928998
- [Result] Seid MH, Rogers R, Dinh Q. The Safety and Tolerability of Ferric Carboxymaltose in Treating Postpartum Women with Iron Dediciency Anemia. American College of Obstetrics & Gynecology District Meeting 2007.
- [Result] Seid MH, Mangione A, Valaoras TG, Anthony LB, Barish CF. Safety Profile of Ferric Carboxymaltose, a New High Dose Intravenous Iron in Patients with Iron Deficiency Anemia. Society for the Advancement of Blood Managment 6th Annual Meeting 2007.
- [Result] Goodnough LT. Treating Postpartum Anemia with Intravenous Ferric Carboxymaltose: a Randomized Controlled Study. Nordic Conference of Obstetrics & Gynecology 2008.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: 1 subject in each group were discontinued from the study prior to dosing due to subject request.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Started | 142 | 147
Completed | 138 | 144
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets | Total
Number analyzed (Participants) | 142 | 147 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 7 | 21
  Between 18 and 65 years | 128 | 140 | 268
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.43 (6.02) | 26.49 (5.55) | 26.45 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 147 | 289
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 142 | 147 | 289

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Classified as a 'Clinical Success'. Clinical Success Was Defined as the Number of Subjects With an Increase in Hemoglobin of >12 g/dL
Time Frame: anytime between baseline and end of study or time to intervention
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Number analyzed (Participants) | 142 | 147
participants | 127 | 98

2. Primary Outcome: Reported Adverse Events
Time Frame: anytime between baseline and end of study or time to intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Ferric Carboxymaltose (FCM) | Ferrous Sulfate Tablets
Serious Adverse Events (participants affected / at risk) | 4/142 | 4/147
Other Adverse Events (participants affected / at risk) | 9/142 | 29/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=142) | Ferrous Sulfate Tablets (N=147)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endometritis (Infections and infestations) | 0 | 2
Pelvic abscess (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=142) | Ferrous Sulfate Tablets (N=147)
Constipation (Gastrointestinal disorders) | 2 | 18
Headache (Nervous system disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less